CLINICAL TRIAL: NCT06980454
Title: A Randomized, Single Intravenous Dose, Parallel Phase I Clinical Study to Compare the Pharmacokinetic Characteristics, Safety, and Immunogenicity of HLX05 Vs. Erbitux® (Cetuximab) in Healthy Adult Male Chinese Subjects
Brief Title: Phase I PK Comparison of HLX05 vs. Erbitux® in Healthy Chinese Males: Safety, Immunogenicity, and Pharmacokinetics
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX05-HV01
Record Dates: First submitted 2025-04-29; First posted 2025-05-20 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Cancer; mCRC
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HLX05 (Experimental)
  Interventions: Drug: HLX05
- US-sourced Erbitux® (Active Comparator)
  Interventions: Drug: US-Erbitux®
- CN-sourced Erbitux® (Active Comparator)
  Interventions: Drug: CN-Erbitux®
- EU-sourced Erbitux® (Active Comparator)
  Interventions: Drug: EU-Erbitux®

INTERVENTIONS:
Drug: HLX05 — A single dose of 250 mg/m2 HLX05 will be given by intravenous drip over 2 h (± 10 min). Antihistamines (e.g., diphenhydramine 20 mg or promethazine 25 mg by intramuscular injection within 30 min prior to dosing) and corticosteroids (e.g., dexamethasone 5 mg by intravenous bolus within 30 min prior to dosing) will be given prior to infusion.
  Arms: HLX05
Drug: EU-Erbitux® — A single dose of 250 mg/m2 EU-Erbitux® injection will be given by intravenous drip over 2 h (± 10 min). Antihistamines (e.g., diphenhydramine 20 mg or promethazine 25 mg by intramuscular injection within 30 min prior to dosing) and corticosteroids (e.g., dexamethasone 5 mg by intravenous bolus within 30 min prior to dosing) will be given prior to infusion.
  Arms: EU-sourced Erbitux®
Drug: US-Erbitux® — A single dose of 250 mg/m2 US-Erbitux® injection will be given by intravenous drip over 2 h (± 10 min). Antihistamines (e.g., diphenhydramine 20 mg or promethazine 25 mg by intramuscular injection within 30 min prior to dosing) and corticosteroids (e.g., dexamethasone 5 mg by intravenous bolus within 30 min prior to dosing) will be given prior to infusion.
  Arms: US-sourced Erbitux®
Drug: CN-Erbitux® — A single dose of 250 mg/m2 US-Erbitux® injection will be given by intravenous drip over 2 h (± 10 min). Antihistamines (e.g., diphenhydramine 20 mg or promethazine 25 mg by intramuscular injection within 30 min prior to dosing) and corticosteroids (e.g., dexamethasone 5 mg by intravenous bolus within 30 min prior to dosing) will be given prior to infusion.
  Arms: CN-sourced Erbitux®

SUMMARY:
This is a randomized, single intravenous dose, parallel study to compare the PK characteristics, safety, tolerability, and immunogenicity of HLX05 vs. Erbitux® (US-, EU-, and CN-sourced) in healthy adult male Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet all the following criteria are allowed to be enrolled:

  1. Males aged 18-50 years (inclusive);
  2. Body mass index (BMI) = body weight (kg)/height2 (m2); BMI between 18.5 and 28.0 (inclusive), and body weight of male subjects ≥ 50 kg;
  3. Subjects without abnormalities or those with abnormalities with no clinical significance in terms of vital signs measurement, physical examination, clinical laboratory tests (hematology, urinalysis, serum chemistry, infectious disease indicators, coagulation function, cardiac markers, alcohol screening, drug screening, etc.), 12-lead ECG examination, chest X-ray, and abdominal B ultrasound;
  4. Subjects who voluntarily take effective contraceptive measures and have no sperm donation plan during the screening period and within 3 months after drug administration, and voluntarily take non-drug contraceptive measures during the trial;

Exclusion Criteria:

* 1. With allergic constitution, or history of food or drug allergy; known history of allergy to any ingredient of the study drug or excipients or monoclonal antibody agents; history of infusion reactions; 2. Subjects with a history of seborrheic dermatitis or other types of dermatitis, rashes, etc., in the past or currently; 3. Subjects with a history of cardiovascular, respiratory, endocrine, hepatic, renal, gastrointestinal, nervous system, or hematological, immunological, psychiatric, metabolic obvious abnormalities, skin diseases, or other significant diseases, and are judged by the investigator as unsuitable for participating in the trial; 4. Those with hereditary bleeding tendency or coagulation disorder, or a history of thrombosis or bleeding disorders; 5. With known or suspected history of keratitis, ulcerative keratitis, or severe dry eye disease;

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 322 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Area under the serum concentration-time curve from time 0 to infinity (AUC0-inf) | up to 29 days

SECONDARY OUTCOMES:
Cmax | up to 29 days
  Maximum serum concentration
Tmax | up to 29 days
  Time to reach maximum serum concentration
CL | up to 29 days
  Total clearance
λz | up to 29 days
  Apparent terminal elimination rate constant

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, Xuzhou, Jiangsu
  - Affiliated Hospital of Xuzhou Medical University, Jiangsu, Xuzhou